CLINICAL TRIAL: NCT02251899
Title: A Disease Management Study Targeted to Reduce Health Care Utilization for Patients With Congestive Heart Failure
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Health Navigator (Other)
Collaborators: Region Stockholm (Other Government); Ostergotland County Council, Sweden (Other); Vastra Gotaland Region (Other Government); Uppsala County Council, Sweden (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HN-AHS-HS-2
Record Dates: First submitted 2014-09-25; First posted 2014-09-29 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: The Focus is to Investigate Effects of a Disease Management Intervention for Patients With Congestive Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Disease-Management intervention (Experimental): Behavioral: Disease-Management intervention The participants in the intervention group receive a nurse-managed disease-management intervention that is regularly delivered by telephone or, when necessary, in person
  Interventions: Behavioral: Disease-Management intervention
- No Intervention: Control arm (No Intervention): Control group not receiving any in

INTERVENTIONS:
Behavioral: Disease-Management intervention — The participants in the intervention group receive a nurse-managed disease-management intervention that is regularly delivered by telephone or, when necessary, in person
  Arms: Disease-Management intervention

SUMMARY:
The aim of this study is to determine whether a nurse-managed telephone-based disease-management intervention can reduce healthcare utilization and improve self-assessed health status in patients with congestive heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ≥1 unplanned inpatient occasion with primary diagnosis of heart failure ( I50) during the last 12 months
* Heart failure grade NYHA II- III
* Accurate heart failure diagnosis
* Living in one of four Swedish counties where the trial is ongoing

Exclusion Criteria:

* Deceased
* In a moribund state
* Significant cognitive loss and therefore cannot provide consent
* Psychosis diagnosis
* Severe hearing impairment
* Language difficulties
* Participants in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2010-01; Primary Completion 2015-12 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Number of hospitalizations | From randomization for up to 2 years
Number of outpatient visits to medical doctor | From randomization for up to 2 years

SECONDARY OUTCOMES:
Mortality | From randomization for up to 2 years
Length of hospital stays | From randomization for up to 2 years
Total health care cost | From randomization for up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Gustaf Edgren, Principal Investigator — gustaf@pheph.se
Locations (1):
- Stockholms Läns Landsting, Stockholm, Sweden

REFERENCES:
- [Result] Reinius P, Johansson M, Fjellner A, Werr J, Ohlen G, Edgren G. A telephone-based case-management intervention reduces healthcare utilization for frequent emergency department visitors. Eur J Emerg Med. 2013 Oct;20(5):327-34. doi: 10.1097/MEJ.0b013e328358bf5a. PMID 22960802